CLINICAL TRIAL: NCT03300921
Title: A Phase Ib Pharmacodynamic Study of Neoadjuvant Paricalcitol in Resectable Pancreatic Cancer
Brief Title: A Phase Ib Pharmacodynamic Study of Neoadjuvant Paricalcitol in Resectable Pancreatic Cancer A Phase Ib Pharmacodynamic Study of Neoadjuvant Paricalcitol in Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Newer research suggested that paricalcitol may be harmful to a subset of pancreatic cancer patients and it is not feasible to subtype patients in the short time frame before surgery
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 26217
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — paricalcitol

STUDY DESIGN:
Intervention Model Description: Arm A: 50mcg IV weekly Arm B: 12mcg PO daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A: 50mcg IV weekly
  Interventions: Drug: Paricalcitol
- Arm B (Experimental): Arm B: 12mcg PO daily
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Product: Paricalcitol
  Dose/Route/Regimen:
  Arm A: 50mcg IV weekly Arm B: 12mcg PO daily

SUMMARY:
The main purpose of this study is to look at the potential effects of paricalcitol (a drug similar to vitamin D) on pancreatic tumors in patients who are planned for surgical removal of their tumor. The study will also look at the safety of paricalcitol prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, apparently resectable, adenocarcinoma of the pancreas at registration.
* Age greater than or equal to 18 years
* Medically fit for surgery in the opinion of the treating surgeon
* Ability to provide written informed consent

Exclusion Criteria:

- Patients who are currently pregnant, planning to become pregnant, or breast-feeding.

Note: women of childbearing potential must agree to use a medically accepted form of birth control including (condoms, diaphragms, cervical cap, an intra-uterine device (IUD), surgical sterility [tubal ligation or a partner that has undergone a vasectomy], or oral contraceptives). OR must agree to completely abstain from intercourse for two weeks before beginning study treatment, during participation in this study, and for 2 weeks after the final study treatment

* Patients with hypercalcemia (blood levels greater than 11.5 mg/dL). Note: In patients with GFR 30-60 mL/min by Cockroft-Gault, blood calcium levels must be 9.5 mg/dL or lower before starting paricalcitol.
* Serum creatinine > 2.5 x ULN OR GFR <30 mL/min by Cockroft-Gault formula . Patients who, in the opinion of the physician, would not be clinically appropriate for receipt of the therapy regimen associated with participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States